CLINICAL TRIAL: NCT01603654
Title: A Randomized Controlled Trial Comparing the Efficacy and Acceptability of Sodium Picosulphate/Magnesium Citrate With Low-volume PEG -Ascorbic Acid as Preparation for Colonoscopy.
Brief Title: Sodium Picosulphate/Magnesium Citrate and Low-volume PEG -Ascorbic Acid as Preparation for Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Dr Gianpiero Manes, MD, Principal investigator, ASST Fatebenefratelli Sacco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Low volume preparations
Record Dates: First submitted 2012-05-17; First posted 2012-05-22 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Colon Cleansing for Colonoscopy
Keywords: Colon preparation; Colonoscopy; Polyethylene glycol; Sodium Picosulphate
MeSH Terms: interventions — MoviPrep

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sodium picosulphate/magnesium citrate (Experimental)
  Interventions: Drug: sodium picosulphate magnesium citrate
- low-volume PEG -ascorbic acid (Active Comparator)
  Interventions: Drug: low-volume PEG -ascorbic acid

INTERVENTIONS:
Drug: sodium picosulphate magnesium citrate — Use of the product in colon cleansing before colonoscopy. Two sachets each containing 10 mg of sodium picosulfate, 3.5 g magnesium oxide and 12.0 g citric acid. The 2 doses are taken diluted in a glass water.
  Other Names: Citrafleet, IBI Lorenzini, Aprilia, Italy
  Arms: sodium picosulphate/magnesium citrate
Drug: low-volume PEG -ascorbic acid — THe product is used as colon cleanser before colonoscopy. It is supplied as a powder for oral use, to be reconstituted with 2 L of water and drunk as a solution. It consists of 100.0 g macrogol 3350 plus electrolytes (7.5 g sodium sulphate, 2.7 g sodium chloride, 1.0 g potassium chloride) and 4.7 g ascorbic acid.
  Other Names: Moviprep, Norgine Ltd, Harefield, UK
  Arms: low-volume PEG -ascorbic acid

SUMMARY:
Adequate bowel cleansing is essential for effective colonoscopy. Acceptance of colon preparation affects the quality of colon cleansing. The study is aimed at comparing the efficacy, safety and acceptability of sodium picosulphate/magnesium citrate (PMC) and low-volume PEG -ascorbic acid (PEG+ASC)in colon cleansing, and to identify predictors of poor bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

* adult outpatients
* aged 18-85 years
* undergoing elective colonoscopy

Exclusion Criteria:

* previous colon resection
* ileus
* intestinal obstruction
* toxic megacolon
* severe heart failure (New York Heart Association [NYHA] Class III or IV)
* acute cardiovascular disease
* uncontrolled arterial hypertension (systolic pressure > 170 mmHg, diastolic pressure > 100 mmHg)
* severe liver failure or ascites
* end-stage renal failure
* phenylketonuria
* glucose-6-phosphate dehydrogenase deficiency. Women were excluded from the study if they were pregnant, breastfeeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of bowel cleansing | Within 24 hrs
  Assessment of quality of colon cleansing at colonoscopy as achieved by the two study products

SECONDARY OUTCOMES:
Safety | In the 24 hours within assumption of study products
  Occurrence of complications related to the intake or the two study products
Tolerability | Within 12 hrs
  Acceptability of the two study products in term of palatability and ease to take the products

CONTACTS AND LOCATIONS:
Overall Officials: Gianpiero Manes, MD, Principal Investigator — Ospedale L. Sacco
Locations (3):
- Italy (3):
  - Ospedale Valduce, Gastroenterologia, Como
  - Ospedale S. Paolo, Milan
  - Ospedale L. Sacco, Endoscopic Unit, Milan